CLINICAL TRIAL: NCT06279273
Title: The Dynamic Network Mechanism for the Risky Decision-making Deficits Among Methamphetamine Dependence Individuals and Its Trans-cranial Current Stimulation
Brief Title: A Study for the Risky Decision-making Deficits Among Methamphetamine Dependence Individuals and Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Wuhan Mental Health Centre (Other); Wuhan Judicial Bureau Hanyang Compulsory Isolated Detoxification Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NZhong-005
Record Dates: First submitted 2024-01-05; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Methamphetamine Use Disorder
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation
- sham tDCS (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Participants were treated for a total of 20 sessions with active or sham stimulation at 2 mA. Each session lasted 20 min at a fixed daytime interval.

SUMMARY:
The risky decision-making deficits is the core feature of the methamphetamine (MA) dependence. Our previous research found that MA dependents have network abnormalities such as decision-making and rewarding. The feedback-related negativity amplitude in the prefrontal central area of MA users becomes smaller and blunted after a loss. Moreover, the neural modulation over the prefrontal cortex showed potent to decrease the craving, and the functional connectivity between frontal cortex and subparietal lobules increases. It suggests that there is a correlation between the decision-making network and the reward network of MA addicts, but there is no real-time observation of the dynamic changes of these brain network activities, so it is difficult to correct the interaction mechanism.

In order to clarify the dynamic brain network mechanism of the risky decision-making deficits among MA dependents, firstly, based on magneto-encephalography source information reconstruction methods, firstly, based on magneto-encephalography source information reconstruction methods, the investigators will observe the sequence and interaction among decision-making network, rewarding network, and emotion network. Besides, the investigators clarify that the trans-cranial current stimulation over prefrontal cortex could improve the speed and intensity of the key network interactions among MA dependents, which could improve risky decision-making and craving. The successful implementation of the study is expected to provide important clues for elucidating the pathological mechanism of risky decision-making deficits in MA dependents and providing a theoretical basis for the treatment of addiction.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of severe MA defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth edition (DSM-5); Normal hearing and vision, or within normal range after correction;

Exclusion Criteria:

Clinical diagnosis of substance use disorder other than an MA or nicotine use disorder defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth edition (DSM-5) in the past 5 years; Suffering from diseases that affect cognitive function (such as cerebrovascular diseases) ; Schizophrenia, bipolar disorder, depression or other Axis I disorder of DSM-V criteria; any contraindication for fMRI scanning.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frontal lobe activation level | Two weeks
  Balloon Analogue Risk Task during fMRI scanning (Philips Ingenia 3.0T MRI).
cue-induced craving | Two weeks,Four weeks
  Craving was assessed by visual analog scales (VAS), with 0 mm being "no craving"and 100 mm representing "most craving ever experienced for methamphetamine ".

SECONDARY OUTCOMES:
Cognitive function | Two weeks
  Chinese version of the CogState Battery was used to assess cognitive function. We selected five tasks: Two back task (working memory), Continuous paired association task (visual spatial working memory), Groton maze learning task (error monitoring), social emotional cognition (social emotional cognition) and Detection task (processing speed) which were displayed on a green screen with standardized instructions before each task beginning.The accuracy in Two back task, social emotional cognition, and the speed in Detection task, and total errors in Continuous paired association task, Groton maze learning task are our focus.

OTHER OUTCOMES:
Attention bias towards methamphetamine | Two weeks
  The Classic Clue Induced Experimental Paradigm is used to evaluate the attention bias towards drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Na Zhong, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China